CLINICAL TRIAL: NCT01908322
Title: SORINT - SORafenib for Treatment of Patients With INTermediate Stage Hepatocellular Carcinoma
Brief Title: Investigating Patient Characteristics of Intermediate Stage Hepatocellular Carcinoma Patients Treated With Nexavar and Their Distribution to Different Treatment Groups as Well as Determining Effectiveness and Safety
Acronym: SORINT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16628
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Intermediate stage; Observational study
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients will be followed-up from start of Nexavar therapy until death or drop out due to any reason or end of study

SUMMARY:
The study aims to investigate patient characteristics of intermediate stage hepatocellular carcinoma patients treated with Nexavar and their distribution to different treatment groups as well as determining efficacy and safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of unresectable intermediate stage hepatocellular carcinoma (BCLC-B) for whom the decision has been taken by the investigator to prescribe Nexavar (the BCLC intermediate stage (BCLC-B) consists of Child-Pugh A and B patients with large/multifocal HCC who do not have cancer related symptoms, macrovascular invasion or extrahepatic spread).

Exclusion Criteria:

- Prior targeted therapy for hepatocellular carcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with intermediate stage hepatocellular carcinoma (BCLC-B) treated with Nexavar according to the local summary of product characteristics. Participants will be recruited from oncological and gastroenterological clinics and practices throughout Germany.
  In this non-interventional observational study, the decision on the duration and dosage of treatment is solely at the discretion of the attending physician.
  The medication is prescribed at regular visits to the investigator's office. Commercially available product will be used to treat the patients.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Distribution of intermediate stage hepatocellular carcinoma (HCC) patients treated with Nexavar to different treatment groups will be evaluated by the relative frequency of patients in each treatment group. | up to 54 months
Characteristics of patients with intermediate stage HCC (BCLC-B) treated with Nexavar will be determined by evaluating demographic data, medical history, previous treatment of HCC, specific concomitant conditions (amongst others). | up to 54 months

SECONDARY OUTCOMES:
Overall Survival is measured as the time interval from start of Nexavar therapy to the date of death, due to any reason. | up to 54 months
Time to progression is defined as the time interval from start of Nexavar therapy to the date of diagnosed progression. | up to 54 months
Progression free survival is measured as the time interval from the start of Nexavar treatment to diagnosed (radiological or clinical) progression or death, whichever comes first. | up to 54 months
Time to treatment failure is defined as the time interval from start of Nexavar therapy to the date of diagnosed progression or permanent discontinuation due to toxicity. | up to 54 months
Duration of Nexavar treatment is measured as the time interval from start of Nexavar therapy to the date of permanent discontinuation of Nexavar therapy (regardless of the reason for discontinuation). | up to 54 months
Tumor status at different visits will be evaluated according to radiological or clinical evaluation. The best overall response will be analyzed providing absolute and relative frequencies of the tumor status categories. | up to 54 months
Further possible prognostic factors will be evaluated. | up to 54 months
Safety variables will be summarized using descriptive statistics based on adverse events collection. | up to 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany